CLINICAL TRIAL: NCT05552092
Title: Optimal Depth for Esophageal Stethoscope for the Monitoring of Core Temperature
Brief Title: Optimal Depth for Esophageal Stethoscope
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chosun University Hospital (Other)
Responsible Party: Principal Investigator, Ki Tae Jung, Professor, Chosun University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ET_Position
Record Dates: First submitted 2022-09-14; First posted 2022-09-23 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Surgery
Keywords: Anatomic Landmarks; Body Temperature; Monitoring, Intraoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): The patients with ASA class 1-2 (20-65 years old) who are undergoing elective surgery with supine or lithotomy position, without position change, scheduled to last more than 90 min.
  Interventions: Device: Esophageal temperature monitoring according to the depth; Other: Anatomical landmark

INTERVENTIONS:
Device: Esophageal temperature monitoring according to the depth — Core temperatures will be measured with a tympanic thermometer as a reference. When the tympanic membrane (TM) temperature is constant after measuring three consecutive times at 10 seconds intervals, the temperature will be assumed as the core body temperature.
  Initially, the esophageal stethoscope (ES) will be inserted to a depth of 45 cm from the incisor. After 30 minutes of monitoring, when the changes in the body temperatures stabilized, initial temperatures of the TM and ES thermistor will be assessed.
  After 5 minutes, ES will be taken out 2 cm back, and the temperatures of each site will be measured when the temperature change of the ES thermistor stabilized below 0.1°C. Eventually, the depth of ES will be changed from 45 to 27 cm with a 2 cm interval, and the temperature at each position will be measured.
Other: Anatomical landmark — For the further evaluation of the optimal insertion depth of GDT, anatomical landmarks such as distance from the cricoid cartilage to the carina (CCD) and distance from the carina to the intervertebral disc between T8 and T9 (CDD) will be measured using an electronic caliper on a preoperative chest X-ray.

SUMMARY:
The purpose of the present study was to evaluate the optimal insertion depth of an esophageal stethoscope with a thermistor for core temperature monitoring.

DETAILED DESCRIPTION:
Monitoring core temperature is crucial for maintaining normothermia during general anesthesia. During anesthesia, an esophageal stethoscope with a thermistor for monitoring esophageal temperature is frequently used.

There are several researches on the depth or position of the esophageal stethoscopes, but there is only limited information (known as about 40-45 cm or T8-T9).

The purpose of the present study was to evaluate the optimal insertion depth of an esophageal stethoscope with a thermistor for core temperature monitoring.

ELIGIBILITY:
Inclusion Criteria:

* The patients with ASA class 1-2 (20-65 years old) who are undergoing elective surgery with supine or lithotomy position, without position change scheduled to last more than 90 min.

Exclusion Criteria:

* anatomical abnormality with the upper airway
* risks of a difficult airway
* abnormal central anatomical structures such as airway, diaphragm, or spine on the chest X-ray
* history of disease or surgery on the stomach or esophagus
* risks of bleeding or coagulopathy on the preoperative laboratory results
* obese patients with BMI over 30
* contraindication to insertion of ES for the surgery
* who did not take a standing chest PA X-ray before surgery
* position change during the surgery
* open chest surgery

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-11-26 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Desired insertion depth of ES thermistor | 1 day
  To evaluate the desired insertion depth, we will assess the accuracy of temperatures of the ES thermistor at each location by estimating the difference between the esophageal temperature using ES thermistor and the core body temperatures of TM.

SECONDARY OUTCOMES:
Correlation analysis | Through study completion, 1 year
  The secondary outcome of the study is to assess the correlation between the characteristics of patients including gender, height, weight, BMI, CCD, or CDD, and the actual insertion depth of the ES which showed the most minor difference in temperature between TM and ES thermistor.
Optimal depth analysis | Through study completion, 1 year
  We will calculate a mathematical model to predict the optimal insertion depth of ES for the esophageal temperature monitoring, and further analysis for the accuracy and correlation will be done.

CONTACTS AND LOCATIONS:
Overall Officials: Ki Tae Jun, M.D., Ph.D., Study Director — Chosun University Hospital
Locations (1):
- Chosun University Hospital, Gwangju, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wang M, Singh A, Qureshi H, Leone A, Mascha EJ, Sessler DI. Optimal Depth for Nasopharyngeal Temperature Probe Positioning. Anesth Analg. 2016 May;122(5):1434-8. doi: 10.1213/ANE.0000000000001213. PMID 26974019